CLINICAL TRIAL: NCT00756613
Title: CSP #465FS - VA Diabetes Trial Long Term Follow-up Study
Brief Title: The VA Diabetes Trial Follow-up Study (VADT-FS)
Acronym: VADT-F
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 465FS
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Diabetes; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 465 VADT participants: The participants had previously participated in the VADT CSP #465 study

SUMMARY:
CSP #465, "Glycemic Control and Complications in Diabetes Mellitus Type 2," was a randomized unblinded clinical trial comparing tight glycemic control to standard glycemic control. Tight glycemic control consisted of giving patients appropriate diabetic medications to lower the patient's HbA1c to around 7%, whereas standard control attempted to lower the patient's HbA1c to between 8% and 9%. The study was conducted at 20 VA medical centers. 1791 patients were randomized over the 2 year accrual period and then followed for an additional 5 years. Follow-up averaged between 5 and 7 years depending upon when the patient was enrolled in the study. Patients were seen on average every three months in the VA Outpatient Clinics. High blood pressure and elevated cholesterol were aggressively treated in patients in both treatment arms. Education regarding diet, exercise, smoking cessation and management of very high and very low glucose was also provided. Data were collected throughout the study on the patients' physical status, adverse and serious adverse events, concomitant medications, and study end points including mortality, heart attack, stroke and surgery to fix the arteries in the heart, legs or neck. The study consisted of broad use of all anti-diabetic treatments commercially available between 2000 and 2008 including oral medications and insulin. Study required medications and all study clinic visits were provided free of the usual VA co-pay. Active clinical follow-up of the sample ended on May 31, 2008. With the end of the clinical trial the patients were transitioned back to usual patient care services, treatment regimens were adjusted where appropriate and future treatment will be dictated by the patient's health and his/her health care provider.

It is important to clarify that with the completion of the active clinical trial and transitioning of patients to this observational trial, all responsibility for the care, treatment and oversight of the study patients will become the responsibility of the patients' Primary Care Physician. The Long Term Follow-up will not collect adverse or serious adverse events, or actively treat or have any "hands-on" care responsibility for the study participants.

The proposed Long Term Follow-up Study will consist of centralized computer database searches and annual survey questionnaires related to quality of life and self-reported events pertinent to the CSP #465 study.

DETAILED DESCRIPTION:
Diabetes mellitus is a major health problem in the U.S., especially in the VA population. The majority of diabetics are Type 2, and they are at risk for microvascular (e.g. eye, kidney) and macrovascular (e.g. cardiovascular) complications. It is probable that many of the macrovascular and microvascular complications potentially prevented by the 5-7 years of good Glycemic control achieved in the VADT (median follow-up 6.25 years) will occur years after completion of the VADT experimental protocol. This follow-up study will provide the opportunity to see if this holds true up to 9 years following the end of 465.

The results will help the VA in evaluating most appropriate treatments and costs of such treatment.

This is a longitudinal observational follow-up study of CSP #465, "Glycemic Control and Complications in Diabetes Mellitus Type 2",the VA Diabetes Trial (VADT) NCT #00032487. The objectives are: 1) to determine the long term effects of intensive glycemic control in type 2 diabetes on major cardiovascular complications (primary outcome), and 2) to determine the long term effects of intensive glycemic control in type 2 diabetes on four secondary outcomes: a) cardiovascular mortality, b) major microvascular complications, c) health-related quality of life, and d) total mortality.

All patients active at the end of VADT will be approached for participation in VADT-FS. The only exclusion reason will be failure to receive consent for participation. Consented VADT-FS patients will be followed until the end of the study unless they withdraw their consent. Patients will be sent a short, standardized self-administered survey annually. Information collected will include: 1) self-reported health status; 2) occurrence of study endpoints; and 3) VA or non-VA outpatient visits, hospitalizations and procedures. A variety of data sources will be searched to verify endpoints. These sources include: 1) VA and non-VA medical records; 2) data from the Centers for Medicare and Medicaid Services (CMS); and 3) VA and US death records. Patients who do not respond to 3 mailed surveys will be contacted by phone.

If still unsuccessful, their designated surrogate will be contacted. Certain endpoints will be adjudicated by the same committee that was utilized by VADT. Endpoints that will be adjudicated will include: 1) cause of death; 2) reason for amputation; and 3) cardiac-related non-VA hospitalizations. Endpoints of interest in this study include: 1) mortality; 2) acute myocardial infarction requiring hospitalization; 3) stroke; 4) new onset congestive heart failure; 5) coronary revascularization; 6) amputation; 7) peripheral revascularization; 8) renal insufficiency; 9) severe visual impairment; and 10) self-reported health status (diabetes-related quality of life).

ELIGIBILITY:
Inclusion Criteria:

* All patients active at the end of VADT will be approached for participation.

Exclusion Criteria:

* The only exclusion criterion will be failure to achieve consent for continued participation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be eligible for the VADT, subjects had to be over 40 years old, have type 2 diabetes and be non-responsive (A1c > 7.5%) to a maximum daily dose of one or more oral agents or on insulin. And to participate in the VADT-FS the participant had to be active in the VADT study.
Sampling Method: Non-Probability Sample
Enrollment: 1044 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Reaven, MD, Study Chair — Phoenix VA Health Care System, Phoenix, AZ; Nicholas Emanuele, MD, Study Chair — Hines VAMC, Hines IL
Locations (2):
- United States (2):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Hines VAMC, Hines IL, Hines, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Azad N, Agrawal L, Emanuele NV, Klein R, Bahn GD, McCarren M, Reaven P, Hayward R, Duckworth W; VADT Study Group. Association of PAI-1 and fibrinogen with diabetic retinopathy in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2014 Feb;37(2):501-6. doi: 10.2337/dc13-1193. Epub 2013 Oct 7. PMID 24101699
- [Result] Azad N, Agrawal L, Emanuele NV, Klein R, Bahn GD, Reaven P; VADT Study Group. Association of blood glucose control and pancreatic reserve with diabetic retinopathy in the Veterans Affairs Diabetes Trial (VADT). Diabetologia. 2014 Jun;57(6):1124-31. doi: 10.1007/s00125-014-3199-7. Epub 2014 Mar 6. PMID 24599110
- [Result] Anderson RJ, Bahn GD, Emanuele NV, Marks JB, Duckworth WC; VADT Study Group. Blood pressure and pulse pressure effects on renal outcomes in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2014 Oct;37(10):2782-8. doi: 10.2337/dc14-0284. Epub 2014 Jul 21. PMID 25048382
- [Result] Hayward RA, Reaven PD, Wiitala WL, Bahn GD, Reda DJ, Ge L, McCarren M, Duckworth WC, Emanuele NV; VADT Investigators. Follow-up of glycemic control and cardiovascular outcomes in type 2 diabetes. N Engl J Med. 2015 Jun 4;372(23):2197-206. doi: 10.1056/NEJMoa1414266. PMID 26039600
- [Result] Saremi A, Schwenke DC, Bahn G, Ge L, Emanuele N, Reaven PD; VADT Investigators. The effect of intensive glucose lowering therapy among major racial/ethnic groups in the Veterans Affairs Diabetes Trial. Metabolism. 2015 Feb;64(2):218-25. doi: 10.1016/j.metabol.2014.10.010. Epub 2014 Oct 17. PMID 25456099
- [Result] Hayward RA, Reaven PD, Emanuele NV; VADT Investigators. Follow-up of Glycemic Control and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2015 Sep 3;373(10):978. doi: 10.1056/NEJMc1508386. No abstract available. PMID 26332555
- [Result] Follow-Up of Glycemic Control and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2015 Jul 9;373(2):198. doi: 10.1056/NEJMx150025. No abstract available. PMID 26154808
- [Result] Azad N, Bahn GD, Emanuele NV, Agrawal L, Ge L, Reda D, Klein R, Reaven PD, Hayward R; VADT Study Group. Association of Blood Glucose Control and Lipids With Diabetic Retinopathy in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2016 May;39(5):816-22. doi: 10.2337/dc15-1897. Epub 2016 Mar 22. PMID 27006510
- [Result] Zimering MB, Knight J, Ge L, Bahn G; VADT Investigators. Predictors of Cognitive Decline in Older Adult Type 2 Diabetes from the Veterans Affairs Diabetes Trial. Front Endocrinol (Lausanne). 2016 Sep 8;7:123. doi: 10.3389/fendo.2016.00123. eCollection 2016. PMID 27660621
- [Result] Herrington WG, Preiss D. Tightening our understanding of intensive glycaemic control. Lancet Diabetes Endocrinol. 2017 Jun;5(6):405-407. doi: 10.1016/S2213-8587(17)30095-5. Epub 2017 Mar 30. No abstract available. PMID 28365412
- [Result] Zoungas S, Arima H, Gerstein HC, Holman RR, Woodward M, Reaven P, Hayward RA, Craven T, Coleman RL, Chalmers J; Collaborators on Trials of Lowering Glucose (CONTROL) group. Effects of intensive glucose control on microvascular outcomes in patients with type 2 diabetes: a meta-analysis of individual participant data from randomised controlled trials. Lancet Diabetes Endocrinol. 2017 Jun;5(6):431-437. doi: 10.1016/S2213-8587(17)30104-3. Epub 2017 Mar 30. PMID 28365411
- [Result] Saremi A, Howell S, Schwenke DC, Bahn G, Beisswenger PJ, Reaven PD; VADT Investigators. Advanced Glycation End Products, Oxidation Products, and the Extent of Atherosclerosis During the VA Diabetes Trial and Follow-up Study. Diabetes Care. 2017 Apr;40(4):591-598. doi: 10.2337/dc16-1875. Epub 2017 Feb 1. PMID 28148544
- [Result] Zhou JJ, Schwenke DC, Bahn G, Reaven P; VADT Investigators. Glycemic Variation and Cardiovascular Risk in the Veterans Affairs Diabetes Trial. Diabetes Care. 2018 Oct;41(10):2187-2194. doi: 10.2337/dc18-0548. Epub 2018 Aug 6. PMID 30082325
- [Result] Zhou JJ, Koska J, Bahn G, Reaven P. Glycaemic variation is a predictor of all-cause mortality in the Veteran Affairs Diabetes Trial. Diab Vasc Dis Res. 2019 Mar;16(2):178-185. doi: 10.1177/1479164119827598. PMID 31014099
- [Result] Davis SN, Duckworth W, Emanuele N, Hayward RA, Wiitala WL, Thottapurathu L, Reda DJ, Reaven PD; Investigators of the Veterans Affairs Diabetes Trial. Effects of Severe Hypoglycemia on Cardiovascular Outcomes and Death in the Veterans Affairs Diabetes Trial. Diabetes Care. 2019 Jan;42(1):157-163. doi: 10.2337/dc18-1144. Epub 2018 Nov 19. PMID 30455335
- [Result] Agrawal L, Azad N, Bahn GD, Ge L, Reaven PD, Hayward RA, Reda DJ, Emanuele NV; VADT Study Group. Long-term follow-up of intensive glycaemic control on renal outcomes in the Veterans Affairs Diabetes Trial (VADT). Diabetologia. 2018 Feb;61(2):295-299. doi: 10.1007/s00125-017-4473-2. Epub 2017 Nov 3. PMID 29101421
- [Result] Reaven PD, Emanuele NV, Wiitala WL, Bahn GD, Reda DJ, McCarren M, Duckworth WC, Hayward RA; VADT Investigators. Intensive Glucose Control in Patients with Type 2 Diabetes - 15-Year Follow-up. N Engl J Med. 2019 Jun 6;380(23):2215-2224. doi: 10.1056/NEJMoa1806802. PMID 31167051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All alive VADT study subjects were approached for participation in the VADT-FS.
Groups:
- 465 VADT Participants - Standard: The participants had previously participated in the VADT trial in the standard of care group.
- 465 VADT Participants - Intensive: The participants had previously participated in the VADT CSP #465 study in the intensive treatment group.
Period: Overall Study
Arm/Group | 465 VADT Participants - Standard | 465 VADT Participants - Intensive
Started | 512 | 532
Completed | 426 | 462
Not Completed | 86 | 70

BASELINE CHARACTERISTICS:
Population: In the original study VADT (NCT00032487) there were 1791 patients, however in the follow-up study there were only 1044 patients consented from the 1791in the VADT study. The patients that did not enter the follow-up study either refused to consent to 465 follow-up study, or died, or withdrew from the original study.
Groups:
- 465 VADT Participants - Standard; 465 VADT Participants -Intensive: The participants had previously participated in the VADT CSP #465 study
- Total: Total of all reporting groups
Arm/Group | 465 VADT Participants - Standard | 465 VADT Participants -Intensive | Total
Number analyzed (Participants) | 512 | 532 | 1044
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 354 | 393 | 747
  >=65 years | 158 | 139 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (8.3) | 59.5 (8.0) | 59.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 498 | 514 | 1012
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 113 | 208
  Not Hispanic or Latino | 417 | 419 | 836
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 9
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 89 | 91 | 180
  White | 409 | 418 | 827
  More than one race | 7 | 11 | 18
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Long Term Effect of Intensive Glycemic Control in Type 2 Diabetes on Major Cardiovascular Complication.
Description: Major CV events (non-fatal MI resulting in hospitalization, non-fatal stroke, new Congestive Heart Failure (CHF), amputation for ischemic diabetic gangrene, or CV-related death).
Time Frame: 15 years
Population: Total number of participants reflect all that participated in the VA Cooperative Studies Program (CSP) #465 study, Glycemic Control and Complications in Diabetes Mellitus Type 2 (VADT) NCT00032487, but censored those who refused to consent to 465 follow-up study or died or withdrew from the study.
Measure: Number; unit: number of events
Groups:
- 465 VADT Participants - Standard: The participants had previously participated in the VADT Cooperative Studies Program (CSP) #465 study in standard treatment group.
- 465 VADT Participants -Intensive: The participants had previously participated in the VADT Cooperative Studies Program (CSP) #465 study in the intensive group.
Arm/Group | 465 VADT Participants - Standard | 465 VADT Participants -Intensive
Number analyzed (Participants) | 899 | 892
number of events | 336 | 325
Statistical Analysis 1: Comparison: 465 VADT Participants - Standard vs 465 VADT Participants -Intensive; To determine the long term effects of intensive glycemic control in type 2 diabetes on major cardiovascular events; Test type: Equivalence — We considered a 20% reduction in primary events to be a reasonable goal of intensive glycemic control over the anticipated 15-year study time period. This effect size was chosen by taking into consideration both the probability of observing an effect of that size given the level of achieved A1c separation, and the perceived value to the patient of this level of benefit relative to the risk and burden of intensive glycemic control; p = 0.24, Regression, Cox; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.78 to 1.06]

2. Secondary Outcome: The Long Term Effects of Intensive Glycemic Control in Type 2 Diabetes on the Secondary Outcome Total Mortality.
Description: The major secondary end-point of cardiovascular (CV) mortality will measure the cause of death (end-stage renal disease, amputation for either ischemic or non-ischemic gangrene, CV-related death, or nonfatal myocardial infarction (MI), stroke, or new congestive heart failure (CHF)) retrieved by the National Death Index (NDI). Survival analysis will analyzed by time of event to death.
Time Frame: 15 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 465 VADT Participants - Standard | 465 VADT Participants -Intensive
Number analyzed (Participants) | 899 | 892
Participants | 366 | 376
Statistical Analysis 1: Comparison: 465 VADT Participants - Standard vs 465 VADT Participants -Intensive; Test type: Equivalence — The equivalence margin is expected 20% reduction for the intensive treatment group compared to the standard treatment group; p = 0.81, Regression, Cox; Cox Proportional Hazard = 1.02, 95% CI 2-sided [0.88 to 1.18]

3. Secondary Outcome: The Long Term Effects of Intensive Glycemic Control in Type 2 Diabetes on the Secondary Outcome Cardiovascular Mortality.
Description: The major secondary end-point of total mortality will measure all deaths with data retrieved from VA Information Resource Center (VIREC) Cooperate Data Warehouse (CDW) . Survival analysis will analyzed by time to death.
Time Frame: 15 years
Population: Total number of participants reflect all that participated in the VA Cooperative Studies Program (CSP) #465 study, Glycemic Control and Complications in Diabetes Mellitus Type 2 (VADT)NCT00032487, but censored those who refused to consent to 465 follow-up study or died or withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 465 VADT Participants - Standard | 465 VADT Participants -Intensive
Number analyzed (Participants) | 899 | 892
Participants | 125 | 118
Statistical Analysis 1: Comparison: 465 VADT Participants - Standard vs 465 VADT Participants -Intensive; Test type: Equivalence — The equivalence margin is 20% reduction of intensive treatment group versus standard treatment group; p = 0.48, Regression, Cox; Cox Proportional Hazard = 0.90, 95% CI 2-sided [0.67 to 1.20]

4. Secondary Outcome: Number of Events on Major Microvascular or Macrovascular Outcome
Description: End-stage renal disease, amputation for either ischemic or non-ischemic gangrene, CV-related death, or nonfatal MI, stroke, or new CHF.
Time Frame: 15 years
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | 465 VADT Participants - Standard | 465 VADT Participants -Intensive
Number analyzed (Participants) | 899 | 892
events | 355 | 342

5. Secondary Outcome: Patients Reported Health Related Quality of Life
Description: Self-reported health status using an instrument adapted for type 2 diabetes mellitus patients from the Diabetes Control and Complications Trial (DCCT) (Duckworth, 1998; Saudek 1996). This survey tool has been used since the inception of the VADT and will be continued in the annual survey. The minimum value is 0 and the maximum value is 100. The higher score is a better outcome.
Time Frame: 9 years
Population: T-test for comparing between the two treatment groups using the average of last two responses of the surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 465 VADT Participants - Standard: The participants had only participated in the VADT Cooperative Studies Program Follow-up #465-F study in standard treatment group.
- 465 VADT Participants -Intensive: The participants had only participated in the VADT Cooperative Studies Program Follow-up #465-F study in the intensive group.
Arm/Group | 465 VADT Participants - Standard | 465 VADT Participants -Intensive
Number analyzed (Participants) | 449 | 470
score on a scale | 62.2 (17.6) | 63.8 (17.2)
Statistical Analysis 1: Comparison: 465 VADT Participants - Standard vs 465 VADT Participants -Intensive; Test type: Equivalence — T-test comparing between the two groups of treatment using the average score of last two surveys; p = 0.172, t-test, 2 sided; Mean Difference (Final Values) = 1.61

ADVERSE EVENTS:
Time Frame: The VA Diabetes Trial Follow-up Study (VADT-FS) has not collected adverse or serious adverse events, is not required to file FDA reports or actively treat or have any "hands-on" care responsibility for the study participants.
Groups:
- EG000: serious and other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | EG000
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT00756613/Prot_SAP_ICF_000.pdf